CLINICAL TRIAL: NCT04715204
Title: Gastrointestinal Tolerance of Under-five Children With Severe Acute Malnutrition to Ready-to-Drink High Energy and Standard Energy Oral Nutrition Supplement Compared to Formula-75/Formula-100
Brief Title: Gastrointestinal Tolerance of Under-five Children With Severe Acute Malnutrition to ONS Compared to F-75/F-100
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: PT. Nutricia Medical Nutrition (Unknown)
Responsible Party: Principal Investigator, Klara Yuliarti, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-04-0406
Record Dates: First submitted 2021-01-12; First posted 2021-01-20 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-12

CONDITIONS: Severe Acute Malnutrition
Keywords: severe acute malnutrition; oral nutrition supplement; Formula-75/Formula-100; Under-five children
MeSH Terms: conditions — Severe Acute Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Formula-75/Formula-100 (Active Comparator): This arm is the control. Formula-75/Formula-100 are the standard formula recommended by WHO to treat severely malnourished children.
  Interventions: Other: Formula-75/Formula-100
- High Energy Oral Nutrition Supplement (Experimental): High energy oral nutrition supplement (ONS) has energy density of 1.5 kcal/ml, with protein-energy ratio of 8.9% and complete micronutrients. It is also named as enteral formula and can be used as a sole source of nutrition. It comes as a ready-to-drink bottled package of 200 mL each. The nutrition fact fulfills the requirement of BPOM (Indonesian Food and Drug Authority) for Special Medical Purpose. The ready-to-drink formula is a safe option to treat severely malnourished patient in terms of hygiene assurance of formula. In Indonesia, many severely malnourished children come from areas with poor access to clean water and proper sanitation. The high energy ONS is beneficial for children who cannot tolerate large volume of feeding.
  Interventions: Other: High Energy Oral Nutrition Supplement
- Standard Energy Oral Nutrition Supplement (Experimental): Standard energy oral nutrition supplement (ONS) has energy density of 1 kcal/ml, with protein-energy ratio of 9.6% and complete micronutrients. It is also named as enteral formula and can be used as a sole source of nutrition. It comes as a ready-to-drink bottled package of 200 mL each. The nutrition fact fulfills the requirement of BPOM (Indonesian Food and Drug Authority) for Special Medical Purpose. The ready-to-drink formula is a safe option to treat severely malnourished patient in terms of hygiene assurance of formula. In Indonesia, many severely malnourished children come from areas with poor access to clean water and proper sanitation.
  Interventions: Other: Standard Energy Oral Nutrition Supplement

INTERVENTIONS:
Other: High Energy Oral Nutrition Supplement — Oral Nutrition Supplement (ONS) or enteral formula is a formula intended to treat individuals who are unable to meet their nutritional requirements through oral diet alone. European Food Safety Authority described ONS as a formula with caloric density >0.9 kcal/mL. Formula with caloric density of >1.2 kcal/mL is categorized as high energy ONS. This intervention has caloric density of 1.5 kcal/mL.
  Other Names: High Energy ONS
  Arms: High Energy Oral Nutrition Supplement
Other: Standard Energy Oral Nutrition Supplement — Oral Nutrition Supplement (ONS) or enteral formula is a formula intended to treat individuals who are unable to meet their nutritional requirements through oral diet alone. European Food Safety Authority described ONS as a formula with caloric density >0.9 kcal/mL. This intervention has caloric density of 1 kcal/mL and it is categorized as standard energy ONS.
  Other Names: Standard Energy ONS
  Arms: Standard Energy Oral Nutrition Supplement
Other: Formula-75/Formula-100 — Formula-75/Formula-100 is a special therapeutic foods to treat children with severe acute malnutrition. WHO designed F75 as a starter formula for stabilization phase with 75 kcal/100 mL, then it is continued with F100 for rehabilitation phase with 100 kcal/100 mL Formula-75 and Formula-100 are made according to recipe from WHO. The ingredients are skimmed milk powder, coconut oil, and sugar. Mineral mix is added, i.e. 2 ml every 100 ml of formula.
  The composition of F-75:
  Skimmed milk 25 g, coconut oil 100 g, sugar 30 g, mineral mix 20 ml, add water to 1000 ml
  The composition of F-100:
  Skimmed milk 80 g, coconut oil 50 g, sugar 60 g, mineral mix 20 ml, add water to 1000 ml
  Other Names: F75/F100
  Arms: Formula-75/Formula-100

SUMMARY:
The primary outcome of the study is to identify gastrointestinal tolerance of under-five children with severe acute malnutrition to ready-to-drink high energy (1.5 kcal/ml) and standard energy (1 kcal/ml) oral nutrition supplement (ONS) compared to Formula-75/Formula-100. The secondary outcomes of the study are weight gain, electrolyte profile and plasma amino acid profile at the beginning and the end of stabilization phase.

In this randomized, controlled trial, 108 patients with severe acute malnutrition will be enrolled. Patients are randomly assigned to 3 groups (Formula-75/Formula-100, high energy ONS, and standard energy ONS) to undergo a two-week treatment. In order to ensure an adequate intake, nasogastric-tube will be placed for home enteral nutrition for at least throughout the two-week study period. Parent or caregiver will be asked to record daily intake, vomit, and defecation score using Bristol stool chart.

DETAILED DESCRIPTION:
The study compares 3 groups of nutrition intervention for severe acute malnourished children aged 6-59 months in terms of gastrointestinal tolerance (primary outcome) and weight gain, electrolyte profile, and amino acid profile (secondary outcomes).

The gastrointestinal tolerance is examined by Bristol stool chart and vomit daily record during 14 days of intervention. Diarrhea is defined according to ESPGHAN, i.e. a decrease in the consistency of stools score (loose or liquid) and an increase in the frequency of evacuations (typically 3 or more in 24 hours). The duration of diarrhea, frequency of diarrhea, and consistency of each stool are recorded.

Vomit will be counted as mean frequency of vomit per day during 14 days intervention. Volume of vomit is recorded. Only vomit due to milk intolerance is counted. Vomit due to irrelevant reasons, such as coughing and crying, will be excluded.

To ensure accurate formula intake, nasogastric tube is placed and patient is admitted for observation for a few days, depending on clinical conditions. Patient is discharged to undergo home enteral nutrition after parent is trained to administer formula and to clean all feeding devices properly. Parents of group F-75/F-100 is trained to make F-75/F-100 at home with hygienic procedure.

The volume of milk intake is recorded daily. Patient is advised not to eat food/drink milk other than the intervention formula.

Protocol for formula advancement is as follows:

* Calorie requirement is calculated by multiplying ideal weight with daily energy requirement (recommended daily allowance, RDA).
* Ideal weight is the median weight for actual height based on WHO growth chart (weight for height/length).
* Height age is the median age corresponding to actual height of patient, based on WHO growth chart (height/length for age)
* The value of RDA is based on height age, which is 110 kcal/day for height age 0-12 months and 100 kcal/kg/day

  1. On the first day: patient is given 50-75% of RDA (recommended daily allowance), the daily volume of formula (F75/standard energy ONS/high energy ONS) will be divided into 8 feeding sessions (every 3 hours). Complete blood count, electrolyte, and amino acid profile will be tested prior to administering formula.
  2. On the second day: patient is given 75-90% of RDA as F75/standard energy ONS/high energy ONS.
  3. On the third day: patient is given 100% of RDA as F100/standard energy ONS/high energy ONS. Serum electrolyte will be tested before administering formula.

Should there be any electrolyte imbalance, the electrolyte level will be corrected according to the clinical guideline.

Weight and height will be measured on the first day and day 14. Head circumference will be measured on the first day.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 12-60 months
* Weight for length/height z score < -3 (WHO 2006)
* Not on nutritional treatment of severe acute malnutrition for the last 1 month

Exclusion Criteria:

* Not willing to take part in this study
* Having diarrhea
* Diagnosed with malignancy or suspected malignancy

Ages: 12 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal tolerance for bowel movement | 14 days
  Frequency of bowel movement per day and description of stool consistency (Bristol stool chart)
Gastrointestinal tolerance for vomit | 14 days
  Frequency of vomit per day and volume of vomit

SECONDARY OUTCOMES:
Weight gain | 14 days
  Weight is measured on day 1 (before intervention) and day 14 (after intervention) in kilogram with 3 decimals. The weight gain is defined as weight on day 14 minus weight on day 1 and will be presented as gram/kg/day.
  Weight on day 1 and day 14 will also be plotted on WHO Growth Chart weight-for-height z-score and the change of weight-for-height z-score will also be measured.
Height gain | 14 days
  Height is measured on day 1 (before intervention) and day 14 (after intervention) in kg with 1 decimals. The height gain is defined as height on day 14 minus height on day 1 and will be presented as centimeter.
  Height on day 1 and day 14 will also be plotted on WHO Growth Chart height-for-age z-score and the change of height-for-age z-score will also be measured.
Prevalence of hypokalemia | Day 1 and day 3
  Prevalence of hypokalemia on day 1 (starting of stabilization phase) and on day 3 (starting of rehabilitation phase). Hypokalemia is defined as serum potassium lower than 3.5 mEq/L.
Prevalence of hypophosphatemia | Day 1 and day 3
  Prevalence of hypophosphatemia on day 1 (starting of stabilization phase) and on day 3 (starting of rehabilitation phase). Hypophosphatemia is defined as serum phophorus inorganic lower than 4 mg/dL (1.29 mmol/L).
Prevalence of hypomagnesemia | Day 1 and day 3
  Prevalence of hypomagnesemia on day 1 (starting of stabilization phase) and on day 3 (starting of rehabilitation phase). Hypomagnesemia is defined as serum magnesium lower than 1.7 mg/dL (0.7 mmol/L).
Changes of plasma amino acid concentration | Day 1 and day 14
  Changes of plasma amino acid concentration between day 1 (beginning of study, stabilization phase) and day 14 (end of the study). Plasma amino acid analysis method is derivatization with butanolic chloride/LC-MS/MS and the measurement result will be presented as µmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Klara Yuliarti, MD, Principal Investigator — Department of Pediatric, Faculty of Medicine, University of Indonesia/ Cipto Mangunkusumo Hospital
Locations (2):
- Indonesia (2):
  - RSUPN Dr. Cipto Mangunkusumo, Jakarta, DKI Jakarta
  - RSUP Fatmawati, Jakarta, DKI Jakarta